CLINICAL TRIAL: NCT01506609
Title: A Randomized, Phase 2 Study of the Efficacy and Tolerability of Veliparib in Combination With Temozolomide or Veliparib in Combination With Carboplatin and Paclitaxel Versus Placebo Plus Carboplatin and Paclitaxel in Subjects With BRCA1 or BRCA2 Mutation and Metastatic Breast Cancer
Brief Title: Study Evaluating Efficacy And Tolerability Of Veliparib in Combination With Temozolomide (TMZ) or In Combination With Carboplatin and Paclitaxel Versus Placebo in Participants With Breast Cancer Gene (BRCA)1 and BRCA2 Mutation and Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-895; 2011-002913-12 (EudraCT Number)
Expanded Access: NCT03123211 (No longer available)
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Breast Cancer
Keywords: PARP; TMZ; Temodal; Carboplatin; veliparib; BRCA2 mutation carrier; Breast cancer; Metastatic breast cancer; temozolomide; BRCA1 mutation carrier; ABT-888; Paclitaxel; Recurrent breast cancer; Temodar; Locally recurrent
MeSH Terms: conditions — Breast Neoplasms | interventions — veliparib; Carboplatin; Temozolomide; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Veliparib with Temozolomide (Experimental): Veliparib 40 mg twice daily (BID) Days 1 through 7 plus TMZ 150 to 200 mg/m^2 QD Days 1 through 5 in each 28-day cycle.
  Interventions: Drug: Veliparib; Drug: Temozolomide
- Placebo with Carboplatin and Paclitaxel (Placebo Comparator): Placebo BID Days 1 through 7 plus carboplatin target area under the curve (mg•min/mL) (AUC) 6 administered on Day 3 of each 21-day cycle and paclitaxel 175 mg/m^2 administered on Day 3 of each 21-day cycle.
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Paclitaxel
- Veliparib with Carboplatin and Paclitaxel (Experimental): Veliparib 80 mg BID Days 1 through 7 plus carboplatin target AUC 6 administered on Day 3 of each 21-day cycle and paclitaxel 175 mg/m^2 administered on Day 3 of each 21-day cycle.
  Interventions: Drug: Veliparib; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo with Carboplatin and Paclitaxel
Drug: Veliparib
  Other Names: ABT-888
  Arms: Veliparib with Carboplatin and Paclitaxel; Veliparib with Temozolomide
Drug: Carboplatin
  Arms: Placebo with Carboplatin and Paclitaxel; Veliparib with Carboplatin and Paclitaxel
Drug: Temozolomide
  Other Names: Temodal
  Arms: Veliparib with Temozolomide
Drug: Paclitaxel
  Other Names: Taxol
  Arms: Placebo with Carboplatin and Paclitaxel; Veliparib with Carboplatin and Paclitaxel

SUMMARY:
The primary objective of the study is to assess the progression-free survival (PFS) of oral veliparib in combination with TMZ or in combination with carboplatin and paclitaxel compared to placebo plus carboplatin and paclitaxel in subjects with BRCA1 or BRCA2 mutation and locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer that is either locally recurrent or metastatic.
* Locally recurrent disease must not be amenable to surgical resection or radiation with curative intent.
* Must have a documented deleterious Breast Cancer Gene BRCA1 or BRCA2 germline mutation.
* If Human Epidermal Growth Factor Receptor (HER2) positive, subjects must have received and progressed on at least one prior standard HER2 directed therapy or the subject must be ineligible to receive anti-HER2 therapy.
* Measurable or non-measurable (but radiologically evaluable) disease by RECIST (Response Evaluation Criteria in Solid Tumors) criteria 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
* Subject must have adequate bone marrow, renal and hepatic function.
* Subject must not be pregnant or plan to conceive a child.

Exclusion Criteria:

* Received anticancer agent(s) or an investigational agent within 21 days prior to C1D1, or radiotherapy within 28 days prior Cycle 1 Day 1.
* More than 2 prior lines of cytotoxic chemotherapy.
* Prior treatment of breast cancer with temozolomide, a platinum agent, or a Poly (ADP ribose) Polymerase (PARP) inhibitor.
* Prior taxane therapy for metastatic breast cancer.
* A history of or evidence of brain metastases or leptomeningeal disease.
* A history of uncontrolled seizure disorder.
* Pre-existing neuropathy from any cause in excess of Grade 1.
* Known history of allergic reaction to cremophor/paclitaxel.
* Clinical significant uncontrolled conditions, active infection, myocardial infarction, stroke, or transient ischemic attack, psychiatric illness/social situations that would limit compliance.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2012-01-23 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (120):
- United States (34):
  - University of Alabama at Birmingham - Main /ID# 62994, Birmingham, Alabama
  - Banner MD Anderson Cancer Ctr /ID# 118695, Gilbert, Arizona
  - University of Arkansas for Medical Sciences /ID# 60750, Little Rock, Arkansas
  - Moore UC San Diego Cancer Center /ID# 60754, La Jolla, California
  - The Angeles Clinic and Researc /ID# 60743, Los Angeles, California
  - Stanford University School of Med /ID# 65488, Stanford, California
  - Cedars-Sinai Medical Center - West Hollywood /ID# 60760, West Hollywood, California
  - Univ of Colorado Cancer Center /ID# 60751, Aurora, Colorado
  - Lynn Cancer Institute, Boca /ID# 60749, Boca Raton, Florida
  - Holy Cross Hospital /ID# 62995, Fort Lauderdale, Florida
  - Moffitt Cancer Center /ID# 60746, Tampa, Florida
  - Florida Cancer Specialists - East /ID# 60762, West Palm Beach, Florida
  - University of Illinois - Chicago /ID# 106175, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 60755, Chicago, Illinois
  - Rush University Medical Center /ID# 65489, Chicago, Illinois
  - Midwestern Regional CTC /ID# 60744, Zion, Illinois
  - Johns Hopkins University /ID# 60759, Baltimore, Maryland
  - Massachusetts General Hospital /ID# 64582, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 93833, Boston, Massachusetts
  - William Beaumont Hospital /ID# 95417, Royal Oak, Michigan
  - Washington University-School of Medicine /ID# 62724, St Louis, Missouri
  - Beth Israel Medical Center /ID# 87993, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 63222, New York, New York
  - Duke University Medical Center /ID# 60747, Durham, North Carolina
  - Penn State University and Milton S. Hershey Medical Center /ID# 62723, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 60753, Philadelphia, Pennsylvania
  - University of Pittsburgh MC /ID# 60758, Pittsburgh, Pennsylvania
  - University of Pittsburgh MC /ID# 65486, Pittsburgh, Pennsylvania
  - Medical University of South Carolina /ID# 60752, Charleston, South Carolina
  - The West Clinic /ID# 65487, Memphis, Tennessee
  - The West Clinic /ID# 94599, Memphis, Tennessee
  - The West Clinic /ID# 94600, Memphis, Tennessee
  - UT Southwestern Medical Center /ID# 60745, Dallas, Texas
  - Houston Methodist Hospital - Scurlock Tower /ID# 60742, Houston, Texas
- Argentina (2):
  - Coiba /Id# 65219, Berazategui, Buenos Aires
  - ISIS Centro Especializado /ID# 65226, Santa Fe
- Australia (8):
  - The Prince of Wales Hospital /ID# 63271, Randwick, New South Wales
  - Southern Medical Day Care Ctr /ID# 63274, Wollongong, New South Wales
  - Mater Misericordiae Limited /ID# 63276, South Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 63280, Adelaide, South Australia
  - Royal Hobart Hospital /ID# 63279, Hobart, Tasmania
  - Peter MacCallum Cancer Ctr /ID# 63272, Melbourne, Victoria
  - Royal Melbourne Hospital /ID# 63278, Parkville, Victoria
  - Mount Hospital /ID# 65262, Perth, Western Australia
- Belgium (6):
  - Cliniques Universitaires Saint Luc /ID# 96135, Woluwe-Saint-Lambert, Brussels Capital
  - Grand Hôpital de Charleroi /ID# 96136, Charleroi, Hainaut
  - AZ St-Jan Brugge-Oostende AV /ID# 107315, Bruges, West-Vlaanderen
  - UZ Antwerp /ID# 96945, Edegem
  - UZ Leuven /ID# 96138, Leuven
  - CHU UCL Namur /ID# 110595, Namur
- Brazil (3):
  - Hospital Bruno Born / Sociedade Beneficencia e Caridade de Lajeado /ID# 65247, Lajeado, Rio Grande do Sul
  - Irmandade da Santa Casa de /ID# 65244, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre /ID# 65242, Porto Alegre, Rio Grande do Sul
- Canada (4):
  - Sunnybrook Health Sciences Ctr /ID# 77373, Toronto, Ontario
  - CHUM - Notre-Dame Hospital /ID# 67862, Montreal, Quebec
  - Jewish General Hospital /ID# 69893, Montreal, Quebec
  - CHUQ-Hospital St. Sacrement /ID# 68902, Québec, Quebec
- Czechia (3):
  - Masarykuv onkologicky ustav /ID# 65170, Brno
  - Palacky University /ID# 63923, Olomouc
  - Vseobecna Fakultni Nemocnice /ID# 65172, Prague
- Denmark (2):
  - Vejle Sygehus /ID# 65173, Vejle, Region Syddanmark
  - Rigshospitalet, Finsen Centre /ID# 67822, Copenhagen
- Finland (2):
  - Docrates Cancer Center /ID# 63924, Helsinki
  - Tampere University Hospital /ID# 102417, Tampere
- France (8):
  - Hopital Universitaire Purpan /ID# 98815, Toulouse, Haute-Garonne
  - Institut de Cancer de l'Ouest /ID# 63927, Saint-Herblain, Loire-Atlantique
  - Centre Leon Berard /ID# 106675, Lyon, Rhone
  - Pays-Basque Ctr Oncology/Radio /ID# 65176, Bayonne
  - Institut Paoli-Calmettes /ID# 65175, Marseille
  - Hopital Rene Huguenin /ID# 65177, Saint-Cloud
  - Centre Paul Strauss /ID# 100275, Strasbourg
  - Institut Curie /ID# 63926, Paris, Île-de-France Region
- Hungary (3):
  - Bajcsy-Zsilinszky Korhaz /ID# 65179, Budapest
  - Debreceni Egyetem Klinikai Kozpont /ID# 65178, Debrecen
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz /ID# 63928, Szolnok
- Israel (8):
  - Rabin Medical Center /ID# 63929, Petakh Tikva, Tel Aviv
  - Soroka University Medical Center /ID# 65180, Beersheba
  - Assaf Harofeh Medical Center /ID# 65181, Be’er Ya‘aqov
  - Rambam Health Care Campus /ID# 63930, Haifa
  - Shaare Zedek Medical Center /ID# 116575, Jerusalem
  - Gastroenterology Institute, Division of Medicine /ID# 63931, Jerusalem
  - Sheba Medical Center /ID# 63932, Ramat Gan
  - Kaplan Medical Center /ID# 63933, Rehovot
- Erasmus Medisch Centrum /ID# 96275, Rotterdam, Netherlands
- Haukeland University Hospital /ID# 67982, Bergen, Hordaland, Norway
- Poland (5):
  - Mrukmed. Lekarz Beata Madej Mruk i Partner /ID# 94975, Rzeszów, Podkarpackie Voivodeship
  - Centrum Onkologii Lukaszczyka /ID# 73393, Bydgoszcz
  - Olsztynski Osrodek Onkologi /ID# 71060, Olsztyn
  - NZOZ Centrum Medyczne HCP /ID# 68102, Poznan
  - Wielkopolskie Centrum Onkologi /ID# 71061, Poznan
- Romania (5):
  - S.C. lanuli Med Consult SRL /ID# 106955, Bucharest
  - lnstitutul Oncologic Trestiore /ID# 96742, Bucharest
  - Spitalul Clinic Judetean de Urgenta /ID# 96741, Cluj-Napoca
  - Inst Oncology Prof. Chiricuta /ID# 96740, Cluj-Napoca
  - Sc Oncolab Srl /Id# 96745, Craiova
- Russia (9):
  - Federal State Budgetary Scientific Institution N.N. Blokhin Russian Cancer Resea /ID# 65263, Moscow, Moscow
  - Chelyabinsk Reg Clin Oncology /ID# 63938, Chelyabinsk
  - State Regional Budgetary Healthcare Institution " Murmansk Regional Oncology Dis /ID# 102415, Murmansk
  - City Clinical Hospital 1 /ID# 102416, Novosibirsk
  - Pyatigorsk Oncology Dispensary /ID# 65264, Pyatigorsk
  - Birch A Healthcare /ID# 65265, Saint Petersburg
  - N.N. Petrov Research Inst Onc /ID# 65269, Saint Petersburg
  - N.N. Petrov Research Inst Onc /ID# 78973, Saint Petersburg
  - Volgograd Reg Onc Disp #3 /ID# 98035, Volzhsky
- Spain (6):
  - Hospital Universitario Vall d'Hebron /ID# 97415, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 97418, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 97417, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 97416, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 97976, Málaga
  - Hospital Clinico Universitario de Valencia /ID# 97975, Valencia
- Sweden (3):
  - Skanes Universitetssjukhus /ID# 96475, Malmo, Skåne County
  - Sahlgrenska University Hosp /ID# 97715, Gothenburg
  - Karolinska Univ Sjukhuset /ID# 98037, Solna
- Ukraine (7):
  - Cherkassy Regional Onc Ctr /ID# 97698, Cherkasy
  - Municipal Non-Profit Enterprise City Clinical Hospital No.4 of Dnipro City Counc /ID# 63940, Dnipro
  - Communal non-profit enterprise Regional Center of Oncology /ID# 97696, Kharkiv
  - Lviv Oncological Regional Therapeutical and Diagnostic Centre /ID# 63941, Lviv
  - Odessa National Medical Univ /ID# 65278, Odesa
  - Poltava Regional Clinical Oncology Centre of Poltava Regional Council /ID# 97697, Poltava
  - Municipal Non-Profit Enterprise of Sumy Regional Council Sumy Regional Clinical /ID# 65280, Sumy

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Han HS, Dieras V, Robson M, Palacova M, Marcom PK, Jager A, Bondarenko I, Citrin D, Campone M, Telli ML, Domchek SM, Friedlander M, Kaufman B, Garber JE, Shparyk Y, Chmielowska E, Jakobsen EH, Kaklamani V, Gradishar W, Ratajczak CK, Nickner C, Qin Q, Qian J, Shepherd SP, Isakoff SJ, Puhalla S. Veliparib with temozolomide or carboplatin/paclitaxel versus placebo with carboplatin/paclitaxel in patients with BRCA1/2 locally recurrent/metastatic breast cancer: randomized phase II study. Ann Oncol. 2018 Jan 1;29(1):154-161. doi: 10.1093/annonc/mdx505. PMID 29045554
- [Derived] Isakoff SJ, Puhalla S, Domchek SM, Friedlander M, Kaufman B, Robson M, Telli ML, Dieras V, Han HS, Garber JE, Johnson EF, Maag D, Qin Q, Giranda VL, Shepherd SP. A randomized Phase II study of veliparib with temozolomide or carboplatin/paclitaxel versus placebo with carboplatin/paclitaxel in BRCA1/2 metastatic breast cancer: design and rationale. Future Oncol. 2017 Feb;13(4):307-320. doi: 10.2217/fon-2016-0412. Epub 2016 Oct 14. PMID 27739325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Under the original protocol, approximately 4 participants were randomized in a 1:1:1 ratio (Group 1) to 1 of the 3 treatment arms (1 participant in veliparib 40 mg twice daily (BID)+temozolomide (TMZ) arm and a total of 3 participants in either the veliparib 80 mg BID+carboplatin+paclitaxel or the placebo BID+carboplatin+paclitaxel arms) at approximately 3 research sites. Participants randomized under the original protocol were in Group 1, and were not included in the primary efficacy analyses.
Pre-assignment Details: Following approval of Amendment 1, the veliparib dose in combination with carboplatin and paclitaxel was increased to 120 mg BID. Participants were randomized 1:1:1 ratio (Group 2) to 1 of the 3 treatment arms (veliparib 40 mg BID+TMZ, veliparib 120 mg BID+carboplatin+paclitaxel, placebo BID+carboplatin+paclitaxel) at approximately 120 research sites. Participants randomized following approval of Amendment 1 were in Group 2 and were included in the primary efficacy analyses.
Groups:
- Group 1 Placebo + Carboplatin/Paclitaxel: Placebo BID Days 1 through 7 plus carboplatin target area under the curve (mg•min/mL) (AUC) 6 administered on Day 3 of each 21-day cycle and paclitaxel 175 mg/m^2 administered on Day 3 of each 21-day cycle.
- Group 1 Veliparib + Carboplatin/Paclitaxel: Veliparib 80 mg BID Days 1 through 7 plus carboplatin target AUC 6 administered on Day 3 of each 21-day cycle and paclitaxel 175 mg/m^2 administered on Day 3 of each 21-day cycle.
- Group 1 Veliparib + TMZ; Group 2 Veliparib + TMZ: Veliparib 40 mg BID Days 1 through 7 plus TMZ 150 to 200 mg/m^2 QD Days 1 through 5 in each 28-day cycle.
- Group 2 Placebo + Carboplatin/Paclitaxel: Placebo BID Days 1 through 7 plus carboplatin carboplatin target AUC 6 administered on Day 3 of each 21-day cycle and paclitaxel 175 mg/m^2 administered on Day 3 of each 21-day cycle.
- Group 2 Veliparib + Carboplatin/Paclitaxel: Veliparib 120 mg BID Days 1 through 7 plus carboplatin target AUC 6 administered on Day 3 of each 21-day cycle and paclitaxel 175 mg/m^2 administered on Day 3 of each 21-day cycle.
Period: Overall Study
Arm/Group | Group 1 Placebo + Carboplatin/Paclitaxel | Group 1 Veliparib + Carboplatin/Paclitaxel | Group 1 Veliparib + TMZ | Group 2 Placebo + Carboplatin/Paclitaxel | Group 2 Veliparib + Carboplatin/Paclitaxel | Group 2 Veliparib + TMZ
Started | 2 | 1 | 1 | 99 | 97 | 94
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 2 | 1 | 1 | 99 | 96 | 94
Not completed — Adverse Event Related to Progression | 0 | 0 | 0 | 3 | 7 | 3
Not completed — Adverse Event Not Related to Progression | 0 | 1 | 0 | 6 | 10 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 9 | 7 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Sponsor Discontinued Study | 0 | 0 | 0 | 2 | 2 | 0
Not completed — Progressive Disease per Protocol | 1 | 0 | 0 | 64 | 57 | 74
Not completed — Other, Not Specified | 0 | 0 | 0 | 10 | 7 | 3
Not completed — Missing / Unknown Reason | 1 | 0 | 1 | 4 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Placebo + Carboplatin/Paclitaxel; Group 2 Placebo + Carboplatin/Paclitaxel: Placebo BID Days 1 through 7 plus carboplatin target AUC 6 administered on Day 3 of each 21-day cycle and paclitaxel 175 mg/m^2 administered on Day 3 of each 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Group 1 Placebo + Carboplatin/Paclitaxel | Group 1 Veliparib + Carboplatin/Paclitaxel | Group 1 Veliparib + TMZ | Group 2 Placebo + Carboplatin/Paclitaxel | Group 2 Veliparib + Carboplatin/Paclitaxel | Group 2 Veliparib + TMZ | Total
Number analyzed (Participants) | 2 | 1 | 1 | 99 | 97 | 94 | 294
Age, Customized [Count of Participants; unit: Participants]
  < 45 years | 2 | 1 | 0 | 47 | 49 | 41 | 140
  45 to 64 years | 0 | 0 | 1 | 49 | 47 | 46 | 143
  >= 65 years | 0 | 0 | 0 | 3 | 1 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 97 | 95 | 92 | 288
  Male | 0 | 0 | 0 | 2 | 2 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 6 | 7 | 5 | 18
  No Ethnicity | 2 | 1 | 1 | 93 | 90 | 89 | 276
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 1 | 93 | 92 | 83 | 272
  Black | 0 | 0 | 0 | 4 | 3 | 10 | 17
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other, Not Specified | 0 | 0 | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the number of months from the date the participant was randomized to the date of radiographic progression as determined by the central imaging center, or to the date of all cause deaths within 63 days of last tumor assessment if disease progression was not reached.
Time Frame: Radiographic evaluation every 9 weeks, clinical evaluation every cycle (data cutoff date: 04 March 2016); maximum duration of follow up for PFS was 34 months.
Population: Group 2: All randomized participants with suspected deleterious or deleterious breast cancer gene (BRCA)1 or BRCA2 mutation determined by sponsor core lab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 2 Placebo + Carboplatin/Paclitaxel | Group 2 Veliparib + Carboplatin/Paclitaxel | Group 2 Veliparib + TMZ
Number analyzed (Participants) | 98 | 95 | 91
months | 12.3 [9.3 to 14.5] | 14.1 [11.5 to 16.2] | 7.4 [5.9 to 8.5]
Statistical Analysis 1: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + Carboplatin/Paclitaxel; Test type: Superiority; p = 0.227, Log Rank; Hazard Ratio (HR) = 0.789, 95% CI 2-sided [0.536 to 1.162]
Statistical Analysis 2: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + TMZ; Test type: Superiority; p = 0.001, Log Rank; Hazard Ratio (HR) = 1.858, 95% CI 2-sided [1.278 to 2.702]

2. Secondary Outcome: Overall Survival (OS)
Description: Time to death for a given participant was defined as the number of months from the day the participant is randomized to the date of the participant's death. All events of death were included, regardless of whether the event occurs while the participant was still taking study drug, or after the participant discontinued study drug. If a participant had not died, then the data will be censored at the date when the participant was last known to be alive.
Time Frame: From Cycle 1 Day 1 until participant's death or 3 years post discontinuation (data cutoff date: 04 March 2016); maximum duration of follow up for OS was 72 months.
Population: Group 2: All randomized participants with suspected deleterious or deleterious BRCA1 or BRCA2 mutation determined by sponsor core lab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 2 Placebo + Carboplatin/Paclitaxel | Group 2 Veliparib + Carboplatin/Paclitaxel | Group 2 Veliparib + TMZ
Number analyzed (Participants) | 98 | 95 | 91
months | 25.4 [18.3 to 32.1] | 28.3 [24.9 to 33.4] | 19.1 [14.3 to 21.3]
Statistical Analysis 1: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + Carboplatin/Paclitaxel; Test type: Superiority; p = 0.368, Log Rank; Hazard Ratio (HR) = 0.848, 95% CI 2-sided [0.590 to 1.218]
Statistical Analysis 2: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + TMZ; Test type: Superiority; p = 0.017, Log Rank; Hazard Ratio (HR) = 1.512, 95% CI 2-sided [1.074 to 2.127]

3. Secondary Outcome: Clinical Benefit Rate (CBR) at Week 18
Description: CBR: percentage of participants who were progression-free at 18 weeks, defined as complete response (CR), partial response (PR), stable disease (SD) or non-CR/non-disease progression (PD) per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1.
  CR: The disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 0 mm. PR: >= 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters (SOD). PD: >= 20% increase in the SOD of target lesions, taking as reference the smallest SOD recorded since the treatment started (baseline or after) or the appearance of >=1 new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD since the treatment started (baseline or after).
Time Frame: Week 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2 Placebo + Carboplatin/Paclitaxel | Group 2 Veliparib + Carboplatin/Paclitaxel | Group 2 Veliparib + TMZ
Number analyzed (Participants) | 98 | 95 | 91
percentage of participants | 87.0 [78.3 to 92.4] | 90.7 [82.2 to 95.2] | 73.0 [62.2 to 81.2]
Statistical Analysis 1: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + Carboplatin/Paclitaxel; Test type: Superiority; p = 0.434, Cochran-Mantel-Haenszel — P-value is from Cochran-Mantel-Haenszel test stratified by estrogen receptor/progesterone receptor status and prior cytotoxic therapy use
Statistical Analysis 2: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + TMZ; Test type: Superiority; p = 0.019, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The objective response rate, defined as percentage of participants with a confirmed CR or PR based on RECIST 1.1 criteria. CR: The disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 0 mm. PR: >= 30% decrease in the sum of diameters of target lesions, taking as reference the baseline SODs.
Time Frame: Radiographic evaluation every 9 weeks, clinical evaluation every cycle (data cutoff date: 04 March 2016); maximum duration of follow up for ORR was 34 months.
Population: Group 2: All randomized participants with suspected deleterious or deleterious BRCA1 or BRCA2 mutation determined by sponsor core lab. Participants with at least 1 measurable lesion at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2 Placebo + Carboplatin/Paclitaxel | Group 2 Veliparib + Carboplatin/Paclitaxel | Group 2 Veliparib + TMZ
Number analyzed (Participants) | 80 | 72 | 70
percentage of participants | 61.3 [49.7 to 71.9] | 77.8 [66.4 to 86.7] | 28.6 [18.4 to 40.6]
Statistical Analysis 1: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + Carboplatin/Paclitaxel; Test type: Superiority; p = 0.027, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + TMZ; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline at Week 18 in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) Sensory Subscale Score
Description: EORTC QLQ-CIPN20 sensory subscale score was calculated following the standard scoring algorithm, transformed to a 0 (low quality of life) to 100 (best quality of life) scale. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 18
Population: Group 2: All randomized participants with suspected deleterious or deleterious BRCA1 or BRCA2 mutation determined by sponsor core lab. Participants with a baseline and post baseline value. Per protocol, this outcome measure was not planned for the Veliparib + TMZ arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 2 Placebo + Carboplatin/Paclitaxel | Group 2 Veliparib + Carboplatin/Paclitaxel
Number analyzed (Participants) | 62 | 69
score on a scale | 13.94 (14.123) | 11.24 (13.954)
Statistical Analysis 1: Comparison: Group 2 Placebo + Carboplatin/Paclitaxel vs Group 2 Veliparib + Carboplatin/Paclitaxel; Test type: Superiority; p = 0.354, ANCOVA — ANCOVA with treatment arm and baseline value as covariate; Least Squares (LS) Mean of Difference = -2.302, 95% CI 2-sided [-7.20 to 2.60], Standard Error of Mean 2.476

ADVERSE EVENTS:
Time Frame: All cause mortality: from enrollment through data cutoff date (04 March 2016); maximum duration of follow up was 72 months. Adverse events (AEs) and serious AEs (SAEs): from first dose of study drug up to 30 days after the last dose of study drug. The median duration of treatment with study drug for Placebo + Carboplatin/Paclitaxel, Veliparib + Carboplatin/Paclitaxel, and Veliparib + TMZ arms were 70 days, 84 days, and 42 days, respectively.
Description: All-Cause Mortality: All randomized participants. AEs/SAEs: As Treated population: all randomized participants who took at least 1 dose of study drug (veliparib/placebo), analyzed by the actual treatment that participant received.
Groups:
- Group 1 Placebo + Carboplatin/Paclitaxel: Placebo BID Days 1 through 7 plus carboplatin carboplatin target AUC 6 administered on Day 3 of each 21-day cycle and paclitaxel 175 mg/m^2 administered on Day 3 of each 21-day cycle.
Arm/Group | Group 1 Placebo + Carboplatin/Paclitaxel | Group 1 Veliparib + Carboplatin/Paclitaxel | Group 1 Veliparib + TMZ | Group 2 Placebo + Carboplatin/Paclitaxel | Group 2 Veliparib + Carboplatin/Paclitaxel | Group 2 Veliparib + TMZ
All-Cause Mortality (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 65/96 | 59/93 | 76/93
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 26/96 | 32/93 | 16/93
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 93/96 | 93/93 | 91/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Placebo + Carboplatin/Paclitaxel (N=2) | Group 1 Veliparib + Carboplatin/Paclitaxel (N=1) | Group 1 Veliparib + TMZ (N=1) | Group 2 Placebo + Carboplatin/Paclitaxel (N=96) | Group 2 Veliparib + Carboplatin/Paclitaxel (N=93) | Group 2 Veliparib + TMZ (N=93)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BETA HAEMOLYTIC STREPTOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EMPYEMA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MASTITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RECALL PHENOMENON (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
CENTRAL NERVOUS SYSTEM LESION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Placebo + Carboplatin/Paclitaxel (N=2) | Group 1 Veliparib + Carboplatin/Paclitaxel (N=1) | Group 1 Veliparib + TMZ (N=1) | Group 2 Placebo + Carboplatin/Paclitaxel (N=96) | Group 2 Veliparib + Carboplatin/Paclitaxel (N=93) | Group 2 Veliparib + TMZ (N=93)
ANAEMIA (Blood and lymphatic system disorders) | 2 (3) | 1 (5) | 0 (0) | 49 (113) | 53 (139) | 26 (52)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (2) | 1 (3) | 0 (0) | 27 (88) | 28 (112) | 16 (55)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 8 (30) | 7 (8)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (13) | 1 (3) | 0 (0) | 70 (373) | 68 (402) | 46 (211)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (5) | 1 (2) | 65 (239) | 66 (312) | 72 (187)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 2 (2) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (8) | 4 (4) | 3 (3)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 2 (3) | 2 (2)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 4 (4) | 4 (6)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 4 (6) | 2 (2)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 12 (15) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 16 (19) | 20 (23) | 15 (24)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (14) | 11 (15) | 7 (14)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 28 (49) | 38 (57) | 38 (57)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 25 (44) | 37 (63) | 19 (27)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 6 (6) | 8 (8)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 15 (23) | 9 (17) | 5 (5)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (7)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 9 (14) | 4 (4)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (3) | 56 (133) | 66 (152) | 69 (166)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 11 (20) | 11 (15) | 5 (6)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 5 (5) | 3 (3)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 22 (36) | 26 (41) | 40 (81)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (29) | 23 (61) | 17 (59)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (8) | 2 (3)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 0 (0) | 57 (141) | 47 (93) | 44 (76)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (8) | 3 (4)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 5 (5)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (2) | 0 (0) | 7 (10) | 9 (10) | 3 (3)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 6 (6) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 14 (18) | 13 (18) | 3 (5)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 14 (20) | 5 (5)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 18 (23) | 15 (16) | 9 (12)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 16 (26) | 18 (24) | 0 (0)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 3 (4) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 12 (18) | 5 (5)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 5 (6) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 20 (28) | 14 (17)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 9 (14) | 12 (13) | 13 (13)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 5 (5)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 5 (10) | 5 (10) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 10 (17) | 13 (20) | 6 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 10 (16) | 10 (12)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (11) | 5 (5)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (12) | 1 (2)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 6 (8) | 4 (5) | 3 (3)
WEIGHT INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 2 (5) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 20 (27) | 22 (30) | 21 (29)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 3 (4) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 6 (7) | 9 (12) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 11 (18) | 17 (21) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 31 (45) | 34 (62) | 14 (18)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 23 (40) | 28 (43) | 24 (32)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 12 (16) | 21 (37) | 6 (6)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 10 (14) | 6 (6)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 4 (5) | 7 (8)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 14 (16) | 8 (8)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 20 (38) | 32 (56) | 8 (9)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 4 (4) | 2 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 23 (39) | 17 (55) | 13 (15)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 18 (28) | 23 (31) | 7 (8)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 12 (34) | 18 (19) | 12 (12)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 31 (41) | 34 (61) | 27 (50)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 4 (4) | 2 (2)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 34 (64) | 42 (60) | 7 (7)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 17 (32) | 17 (24) | 4 (4)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 22 (47) | 31 (64) | 4 (5)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 10 (13) | 5 (9)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 7 (8) | 4 (4)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 23 (26) | 14 (16) | 20 (21)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5) | 1 (2)
BREAST PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (23) | 21 (27) | 13 (23)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 22 (28) | 14 (16) | 8 (11)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 7 (8) | 3 (8)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (8) | 2 (2)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 8 (10) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 55 (69) | 61 (79) | 10 (13)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 6 (7) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 12 (16) | 9 (9)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 17 (23) | 7 (10) | 5 (7)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (4) | 6 (10)
HOT FLUSH (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 8 (12) | 14 (22) | 11 (13)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 2 (2) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT01506609/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT01506609/SAP_001.pdf